CLINICAL TRIAL: NCT06052566
Title: An Open-Label, Single-Dose Study to Evaluate the Pharmacokinetics of Efinopegdutide (MK-6024) in Participants With Moderate and Severe Hepatic Impairment
Brief Title: A Study of Efinopegdutide in Participants With Hepatic Impairment (MK-6024-014)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6024-014; MK-6024-014 (Registry Identifier: MSD)
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Results first posted 2025-10-22 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Non-alcoholic Steatohepatitis; Hepatic Impairment
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Efinopegdutide in Participants with Moderate Hepatic Impairment (Experimental): Participants with moderate hepatic impairment received a single 7 mg dose of efinopegdutide 14 mg/ml by subcutaneous (SC) injection.
  Interventions: Drug: Efinopegdutide
- Efinopegdutide in Participants with Severe Hepatic Impairment (Experimental): Participants with severe hepatic impairment received a single 7 mg dose of efinopegdutide 14 mg/ml by SC injection.
  Interventions: Drug: Efinopegdutide
- Efinopegdutide in Healthy-Matched Control Group (Experimental): Healthy matched participants received a single 7 mg dose of efinopegdutide 14 mg/ml by SC injection.
  Interventions: Drug: Efinopegdutide

INTERVENTIONS:
Drug: Efinopegdutide — Subcutaneous injection administered at a dose of 7 mg
  Other Names: MK-6024; HM12525A; JNJ-64565111

SUMMARY:
The purpose of this study was to evaluate the pharmacokinetics of efinopegdutide in participants with hepatic impairment compared to healthy participants, and to examine the safety and tolerability of efinopegdutide.

ELIGIBILITY:
The main inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria:

* A participant assigned female at birth is eligible to participate if not pregnant or breastfeeding, is not a participant of childbearing potential (POCBP), or is a POCBP and agrees to follow contraceptive guidance during the study intervention period and for at least 35 days after the last dose of study intervention.
* For participants with moderate or severe hepatic impairment: Have a diagnosis of chronic (>6 months), stable, hepatic impairment with features of cirrhosis due to any etiology (stability of hepatic disease should correspond to no acute episodes of illness within the previous 2 months due to deterioration in hepatic function).

Exclusion Criteria:

* History of cancer (malignancy).
* Had major surgery and/or donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the prestudy (screening) visit.
* Participants with moderate or severe hepatic impairment who are positive for human immunodeficiency virus (HIV)-1 or HIV-2 at the prestudy (screening) visit.
* Participants with moderate or severe hepatic impairment who received antiviral and/or immune modulating therapy for hepatitis B virus (HBV) or hepatitis C virus (HCV) within 90 days prior to study start.
* Healthy participants who are unable to refrain from or anticipate the use of any medication, including prescription and nonprescription drugs or herbal remedies beginning approximately 2 weeks (or 5 half-lives) prior to administration of the initial dose of study intervention, throughout the study (including washout intervals between treatment periods), until the poststudy visit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-11-21 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (4):
- United States (4):
  - Clinical Pharmacology of Miami ( Site 0005), Miami, Florida
  - Advanced Pharma CR, LLC ( Site 0001), Miami, Florida
  - Genesis Clinical Research, LLC ( Site 0006), Tampa, Florida
  - American Research Corporation ( Site 0002), San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Efinopegdutide in Participants With Moderate Hepatic Impairment | Efinopegdutide in Participants With Severe Hepatic Impairment | Efinopegdutide in Healthy-Matched Control Group
Started | 8 | 8 | 6
Completed | 8 | 8 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Efinopegdutide in Participants With Moderate Hepatic Impairment | Efinopegdutide in Participants With Severe Hepatic Impairment | Efinopegdutide in Healthy-Matched Control Group | Total
Number analyzed (Participants) | 8 | 8 | 6 | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.5 (9.5) | 48.5 (10.5) | 56.2 (7.1) | 53.9 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 3 | 7
  Male | 4 | 8 | 3 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 6 | 19
  Not Hispanic or Latino | 2 | 1 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 8 | 8 | 5 | 21
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time 0 to Infinity (AUC0-inf) of Efinopegdutide
Description: Blood samples collected at multiple timepoints post-dose were used to determine the AUC0-inf.
Time Frame: At pre-specified timepoints on Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 11, Day 14, Day 21, and Day 35
Population: All participants who complied with the protocol sufficiently to ensure that generated data will be likely to exhibit the effects of treatment, according to the underlying scientific model.
Measure: Geometric Mean (95% Confidence Interval); unit: hr*μg/mL
Arm/Group | Efinopegdutide in Participants With Moderate Hepatic Impairment | Efinopegdutide in Participants With Severe Hepatic Impairment | Efinopegdutide in Healthy-Matched Control Group
Number analyzed (Participants) | 6 | 7 | 6
hr*μg/mL | 143 [120 to 169] | 152 [106 to 219] | 146 [81.8 to 262]
Statistical Analysis 1: Comparison: Efinopegdutide in Participants With Moderate Hepatic Impairment vs Efinopegdutide in Healthy-Matched Control Group; Test type: Other; Geometric Mean Ratio = 0.97, 90% CI 2-sided [0.61 to 1.54]
Statistical Analysis 2: Comparison: Efinopegdutide in Participants With Severe Hepatic Impairment vs Efinopegdutide in Healthy-Matched Control Group; Test type: Other; Geometric Mean Ratio = 1.04, 90% CI 2-sided [0.63 to 1.71]

2. Primary Outcome: Area Under the Curve From Time 0 to Last Sampling Time (AUC0-last) of Efinopegdutide
Description: Blood samples collected at multiple timepoints post-dose were used to determine the AUC0-last.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: hr*μg/mL
Arm/Group | Efinopegdutide in Participants With Moderate Hepatic Impairment | Efinopegdutide in Participants With Severe Hepatic Impairment | Efinopegdutide in Healthy-Matched Control Group
Number analyzed (Participants) | 7 | 8 | 6
hr*μg/mL | 133 [113 to 156] | 125 [80.8 to 193] | 134 [70.2 to 255]
Statistical Analysis 1: Comparison: Efinopegdutide in Participants With Moderate Hepatic Impairment vs Efinopegdutide in Healthy-Matched Control Group; Test type: Other; Geometric Mean Ratio = 0.99, 90% CI 2-sided [0.60 to 1.65]
Statistical Analysis 2: Comparison: Efinopegdutide in Participants With Severe Hepatic Impairment vs Efinopegdutide in Healthy-Matched Control Group; Test type: Other; Geometric Mean Ratio = 0.93, 90% CI 2-sided [0.53 to 1.65]

3. Primary Outcome: Maximum Plasma Concentration (Cmax) of Efinopegdutide
Description: Blood samples collected at multiple timepoints post-dose were used to determine the Cmax.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Efinopegdutide in Participants With Moderate Hepatic Impairment | Efinopegdutide in Participants With Severe Hepatic Impairment | Efinopegdutide in Healthy-Matched Control Group
Number analyzed (Participants) | 7 | 8 | 6
μg/mL | 0.348 [0.282 to 0.429] | 0.404 [0.242 to 0.675] | 0.474 [0.253 to 0.890]
Statistical Analysis 1: Comparison: Efinopegdutide in Participants With Moderate Hepatic Impairment vs Efinopegdutide in Healthy-Matched Control Group; Test type: Other; Geometric Mean Ratio = 0.73, 90% CI 2-sided [0.44 to 1.21]
Statistical Analysis 2: Comparison: Efinopegdutide in Participants With Severe Hepatic Impairment vs Efinopegdutide in Healthy-Matched Control Group; Test type: Other; Geometric Mean Ratio = 0.85, 90% CI 2-sided [0.47 to 1.53]

4. Primary Outcome: Time to Maximum Concentration (Tmax) of Efinopegdutide
Description: Blood samples collected at multiple timepoints post-dose were used to determine the Tmax of efinopegdutide.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | Efinopegdutide in Participants With Moderate Hepatic Impairment | Efinopegdutide in Participants With Severe Hepatic Impairment | Efinopegdutide in Healthy-Matched Control Group
Number analyzed (Participants) | 7 | 8 | 6
hour | 120.00 [96.00 to 310.93] | 72.04 [24.00 to 144.00] | 83.78 [48.00 to 167.25]

5. Primary Outcome: Apparent Terminal Half-life (t/12) of Efinopegdutide
Description: Blood samples collected at multiple timepoints post-dose were used to determine the t1/2.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Efinopegdutide in Participants With Moderate Hepatic Impairment | Efinopegdutide in Participants With Severe Hepatic Impairment | Efinopegdutide in Healthy-Matched Control Group
Number analyzed (Participants) | 6 | 7 | 6
hour | 146 (13.5) | 149 (26.0) | 115 (32.3)

6. Primary Outcome: Apparent Total Clearance (CL/F) of Efinopegdutide
Description: Blood samples collected at multiple timepoints post-dose were used to determine the CL/F.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Efinopegdutide in Participants With Moderate Hepatic Impairment | Efinopegdutide in Participants With Severe Hepatic Impairment | Efinopegdutide in Healthy-Matched Control Group
Number analyzed (Participants) | 6 | 7 | 6
L/hr | 0.0491 (16.5) | 0.0460 (40.8) | 0.0478 (60.0)

7. Primary Outcome: Apparent Volume of Distribution (Vz/F) of Efinopegdutide
Description: Blood samples collected at multiple timepoints post-dose were used to determine the Vz/F.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Efinopegdutide in Participants With Moderate Hepatic Impairment | Efinopegdutide in Participants With Severe Hepatic Impairment | Efinopegdutide in Healthy-Matched Control Group
Number analyzed (Participants) | 6 | 7 | 6
Liters | 10.3 (17.9) | 9.88 (57.8) | 7.94 (91.7)

8. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE is defined as any untoward medical occurrence associated with the use of a drug in a participant, whether or not considered drug related. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product and does not imply any judgment about causality.
Time Frame: Up to 35 days
Population: All participants who received at least 1 dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Efinopegdutide in Participants With Moderate Hepatic Impairment | Efinopegdutide in Participants With Severe Hepatic Impairment | Efinopegdutide in Healthy-Matched Control Group
Number analyzed (Participants) | 8 | 8 | 6
Participants | 3 | 4 | 4

9. Secondary Outcome: Number of Participants Who Discontinued Study Intervention Due to an AE
Description: as for outcome 8
Time Frame: Up to 35 days
Population: All participants who received at least 1 dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Efinopegdutide in Participants With Moderate Hepatic Impairment | Efinopegdutide in Participants With Severe Hepatic Impairment | Efinopegdutide in Healthy-Matched Control Group
Number analyzed (Participants) | 8 | 8 | 6
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 35 days
Description: All-Cause Mortality is reported for all randomized participants. Serious adverse events and other adverse events are reported for all participants who received treatment.
Arm/Group | Efinopegdutide in Participants With Moderate Hepatic Impairment | Efinopegdutide in Participants With Severe Hepatic Impairment | Efinopegdutide in Healthy-Matched Control Group
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 2/8 | 4/8 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Efinopegdutide in Participants With Moderate Hepatic Impairment (N=8) | Efinopegdutide in Participants With Severe Hepatic Impairment (N=8) | Efinopegdutide in Healthy-Matched Control Group (N=6)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Efinopegdutide in Participants With Moderate Hepatic Impairment (N=8) | Efinopegdutide in Participants With Severe Hepatic Impairment (N=8) | Efinopegdutide in Healthy-Matched Control Group (N=6)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-31): https://cdn.clinicaltrials.gov/large-docs/66/NCT06052566/Prot_SAP_000.pdf